CLINICAL TRIAL: NCT00412373
Title: A Randomized, Double-blind, Placebo-controlled, Parallel- Group Study to Evaluate the Efficacy and Safety of Flexible-dose Paliperidone ER in the Treatment of Patients With Schizoaffective Disorder.
Brief Title: Evaluation of Effectiveness and Safety of Flexible-dose Paliperidone Extended Release in Patients With Schizoaffective Disorder.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR013099; R076477SCA3002
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Results first posted 2009-12-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Schizoaffective Disorder; Psychotic Disorder
Keywords: Schizoaffective Disorder; antipsychotic; paliperidone; placebo
MeSH Terms: conditions — Psychotic Disorders | interventions — Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 001 (Experimental): Paliperidone ER (3-12mg/day in 3 mg/day increments for 6 weeks)
  Interventions: Drug: Paliperidone ER
- 003 (Experimental): Paliperidone ER (3-12mg/day in 3 mg/day increments for 6 weeks)
  Interventions: Drug: Paliperidone ER
- 002 (Placebo Comparator): Placebo for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — for 6 weeks
  Arms: 002
Drug: Paliperidone ER — (3-12mg/day in 3 mg/day increments for 6 weeks)
  Arms: 003
Drug: Paliperidone ER — (3-12mg/day in 3 mg/day increments for 6 weeks)
  Arms: 001

SUMMARY:
The purpose of this study is to measure the effectiveness and assess the safety of different dosages (from 3 mg/day to 12 mg/day) of the antipsychotic paliperidone extended-release (ER) in patients who are experiencing an acute episode of schizoaffective disorder.

DETAILED DESCRIPTION:
Schizophrenia and schizoaffective disorder are closely related in terms of symptoms, coexisting conditions, and genetic risk. In previous studies in patients with schizophrenia, treatment with paliperidone extended-release (ER) improved psychotic symptoms, as well as mood symptoms evaluated by anxiety/depression and hostility/excitement Positive and Negative Symptoms of Schizophrenia (PANSS) factor scores. Therefore, paliperidone ER may also be effective in treating symptoms of schizoaffective disorder. Paliperidone's limited potential for drug-drug interaction is particularly important in this patient population, in which multiple drug therapy is relatively common. This multicenter, double-blind (neither the patient nor the physician knows whether drug or placebo is being taken, or at what dosage), randomized (patients are assigned different treatments based on chance), placebo-controlled, parallel-group study is designed to examine the effectiveness and safety of paliperidone ER in adult patients with schizoaffective disorder who are experiencing an acute episode of this disorder. Patients in the study will be randomly assigned to 1 of 2 groups to receive 6 weeks of oral treatment with flexible dosages of paliperidone ER (3-12 mg/day) or with placebo. The primary efficacy outcome will be the change from baseline to Week 6, or the last post-randomization assessment during double-blind treatment (endpoint), in the PANSS total score. Safety will be assessed by monitoring adverse events, clinical laboratory testing, pregnancy testing, vital signs measurements, physical examination, administration of a 12-lead ECG, movement disorders side effect scales, and the InterSePT Scale for Suicidal Thinking. Patients may also choose to participate in a pharmacogenomic (DNA) analysis. The primary study hypothesis is that flexible-dose paliperidone ER is better than placebo on the change from baseline in the PANSS total score in acutely ill patients with schizoaffective disorder. Patients will receive study drug by mouth for a total of 43 days. Beginning on Day 1, patients will take either placebo or paliperidone ER 6 mg/day. After day 4, dosages may be adjusted, at defined intervals, to a dosage between 3 mg/day and 12 mg/day, inclusive.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual - Fourth Edition (DSM-IV) diagnosis of schizoaffective disorder
* A total Positive and Negative Symptoms of Schizophrenia (PANSS) score of >= 60
* A score of >= 16 on Young Mania Rating Scale (YMRS) or a score of >= 16 on the Hamilton Depression Rating Scale (HAM-D 21)

Exclusion Criteria:

* A primary active mental illness diagnosis other than schizoaffective disorder
* Patients with first episode psychosis
* Active substance dependence within previous 6 months
* Treatment with clozapine within 6 months of randomization
* A history of treatment resistance, defined by failure to respond to 2 adequate trials of antipsychotic medication
* Pregnancy, breast-feeding, or planning to become pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2006-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (44):
- United States (15):
  - Cerritos, California
  - Costa Mesa, California
  - Garden Grove, California
  - Huntington Beach, California
  - Pico Rivera, California
  - San Diego, California
  - Aventura, Florida
  - Hollywood, Florida
  - Kissimmee, Florida
  - Leesburg, Florida
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Austin, Texas
  - Irving, Texas
- India (8):
  - Ahmedabad
  - Ahmedibad
  - Aurangabad
  - Chennai
  - Delhi
  - Kanpur Uttarpradeh
  - Pune
  - Vadadora
- Malaysia (4):
  - Ipoh
  - Kota Kinabalu
  - Kuala Lumpur
  - Kuching
- Philippines (4):
  - Davao City
  - Mandaluyong
  - Manila
  - Pasig National Capitol Region
- Romania (6):
  - Arad
  - Bucharest
  - Câmpina
  - Com Gura Ocnitei
  - Iași
  - Piteşti
- South Korea (7):
  - Daegu
  - Gyeonggi-do
  - Inchun
  - Jeonju
  - Kwangiu
  - Pusan
  - Seoul

REFERENCES:
- [Derived] Alphs L, Fu DJ, Turkoz I. Paliperidone for the treatment of schizoaffective disorder. Expert Opin Pharmacother. 2016;17(6):871-83. doi: 10.1517/14656566.2016.1161029. Epub 2016 Mar 24. PMID 26934062
- See also: Evaluation of Effectiveness and Safety of Flexible-Dose Paliperidone Extended Release in Patients With Schizoaffective Disorder. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=67&filename=CR013099_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 391 subjects were enrolled in the study. There were 80 screen fails (did not meet inclusion/exclusion criteria). 311 subjects were randomized. 309 subjects were included in the Safety Analysis Set (randomized and took at least one dose of study drug). 304 subjects were included in the Intent-to-Treat analysis set (had baseline/postbase PANSS).
Groups:
- Placebo: A placebo control was used to establish the frequency and magnitude of changes in clinical endpoints that could occur in the absence of active treatment.
- Paliperidone Extended-Release (ER): Paliperidone (9-hydroxy-risperidone, R076477) is an atypical antipsychotic agent approved for the treatment of schizophrenia and is in development for the treatment of bipolar disorder and schizoaffective disorder. Paliperidone is a monoaminergic antagonist that exhibits the characteristic dopamine type 2 (D2) and serotonin (5-hydroxytryptamine [5-HT]) type 2A (5HT2A) antagonism of the newer, or second-generation, antipsychotic drugs. Paliperidone is available in an oral formulation using extended-release (ER).
Period: Overall Study
Arm/Group | Placebo | Paliperidone Extended-Release (ER)
Started | 93 (Number of Subjects in Intent-to-Treat Analysis Set.) | 211 (Number of Subjects Intent-to-Treat Analysis Set.)
Completed | 52 (Number of Subjects Who Completed Double-Blind Treatment.) | 134 (Number of Subjects Who Completed Double-Blind Treatment..)
Not Completed | 41 | 77
Not completed — Adverse Event | 8 | 13
Not completed — Lack of Efficacy | 16 | 22
Not completed — Lost to Follow-up | 7 | 13
Not completed — Withdrawal by Subject | 8 | 27
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Paliperidone Extended-Release (ER) | Total
Number analyzed (Participants) | 93 | 211 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] — The Intent-to-Treat (ITT) analysis set included all randomly assigned subjects who received at least 1 dose of study medication (or any portion of a dose) and had both baseline and at least 1 postbaseline PANSS assessment. ITT for Placebo is 93 subjects and for PALI ER is 211 subjects.
  years | 37.3 (9.4) | 37.7 (9.1) | 37.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Intent-to-Treat (ITT) analysis set. ITT for Placebo is 93 subjects and for PALI ER is 211 subjects.
  Participants
    Female | 39 | 95 | 134
    Male | 54 | 116 | 170
Race (NIH/OMB) [Count of Participants; unit: Participants] — Intent-to-Treat (ITT) analysis set. ITT for Placebo is 93 subjects and for PALI ER is 211 subjects.
  Participants
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 29 | 61 | 90
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 17 | 38 | 55
    White | 47 | 109 | 156
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Symptoms of Schizophrenia (PANSS) Total Score at Baseline.
Description: The PANSS is a 30-item scale (range 30-210) designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items. Higher scores indicate worsening.
Time Frame: Baseline
Population: The Intent-to-Treat population included all randomly assigned subjects who received at least 1 dose of study medication (or any portion of a dose) and had both baseline and at least 1 postbaseline PANSS assessment.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Paliperidone Extended-Release (ER)
Number analyzed (Participants) | 93 | 211
points on a scale | 91.7 (12.1) | 92.3 (13.5)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended-Release (ER); Test type: Superiority or Other; p = 0.774, ANOVA; P-value based on the actual value and was from an ANOVA model with fixed effects for treatment, concomitant medication stratum, and country; LS Mean Difference = 0.5, 95% CI [-2.7 to 3.7], Standard Error of Mean 1.6 — Paliperidone Extended Release (ER) - Placebo on the Actual Score

2. Primary Outcome: Positive and Negative Symptoms of Schizophrenia (PANSS) Total Score - Change From Baseline to Week 6 Last Observation Carried Forward (LOCF) End Point.
Description: as for outcome 1
Time Frame: The primary efficacy endpoint was the change from baseline to week 6 or the last post-randomization assessment during double-blind treatment in the PANSS total score.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Paliperidone Extended-Release (ER)
Number analyzed (Participants) | 93 | 211
points on a scale | -10.8 (18.7) | -20.0 (18.9)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended-Release (ER); Test type: Superiority or Other; p < 0.001, ANCOVA; P-values are from an ANCOVA model with fixed effects for treatment, concomitant medication stratum, and country, and baseline value as a covariate; LS Mean Difference = -9.4, 95% CI [-13.8 to -4.9], Standard Error of Mean 2.3 — Paliperidone Extended Release (ER) - Placebo on the Change Scores

3. Secondary Outcome: Positive and Negative Symptoms of Schizophrenia (PANSS) Positive Subscale Score - Change From Baseline to Week 6 Last Observation Carried Forward (LOCF) End Point.
Description: Positive Syndrome Scale (range 7-49): Sum of scores for items 1-7 in positive subscale: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. Higher scores indicate worsening.
Time Frame: Change from baseline to Week 6 or the last post-randomization assessment during double-blind treatment
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Paliperidone Extended-Release (ER)
Number analyzed (Participants) | 93 | 211
points on a scale | -4.6 (6.3) | -7.3 (6.9)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended-Release (ER); Test type: Superiority or Other; p < 0.001, ANCOVA; P-value is from an ANCOVA model with fixed effects for treatment, concomitant medication stratum, and country, and with baseline value as a covariate; LS Means Difference = -2.8, 95% CI [-4.4 to -1.2], Standard Error of Mean 0.8 — Paliperidone Extended Release (ER) - Placebo on the Change Scores

4. Secondary Outcome: Positive and Negative Symptoms of Schizophrenia (PANSS) Negative Subscale Score - Change From Baseline to Week 6 Last Observation Carried Forward (LOCF) End Point.
Description: Negative Syndrome Scale (range 7-49): Sum of scores for items 1-7 in negative subscale: blunted effect, emotional withdrawal, poor rapport, passive apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, and stereotyped thinking. Higher scores indicate worsening.
Time Frame: Change from baseline to Week 6 or the last post-randomization assessment during double-blind treatment
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Paliperidone Extended-Release (ER)
Number analyzed (Participants) | 93 | 211
points on a scale | -1.1 (5.5) | -3.0 (4.9)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended-Release (ER); Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Means Difference = -2.0, 95% CI [-3.1 to -0.8], Standard Error of Mean 0.6 — Paliperidone Extended Release (ER) - Placebo on the Change Scores

5. Secondary Outcome: Positive and Negative Symptoms of Schizophrenia (PANSS) General Psychopathology Subscale Score - Change From Baseline to Week 6 Last Observation Carried Forward (LOCF) End Point.
Description: General Psychopathology (range 16-112): Sum of scores for somatic concern, anxiety, guilt feelings, tension, mannerisms/posturing, depression, motor retardation, uncooperativeness, unusual thought content, disoriented, poor attention, lack of judgment/insight, disturbance of volition, poor impulse control, preoccupation, and active social avoidance. Higher scores indicate worsening.
Time Frame: Change from baseline to Week 6 or the last post-randomization assessment during double-blind treatment
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Paliperidone Extended-Release (ER)
Number analyzed (Participants) | 93 | 211
points on a scale | -5.2 (9.4) | -9.7 (9.9)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended-Release (ER); Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Means Difference = -4.5, 95% CI [-6.8 to -2.3], Standard Error of Mean 1.2 — Paliperidone Extended Release (ER) - Placebo on the Change Scores

6. Secondary Outcome: Positive and Negative Symptoms of Schizophrenia (PANSS) Positive Factor Score - Change From Baseline to Week 6 Last Observation Carried Forward (LOCF) End Point.
Description: Positive PANSS Factor Score (range 8-56): Sum of scores for items 1, 3, 5, and 6 in positive subscale: delusions, hallucinatory behavior, grandiosity, suspiciousness; item 7 in negative subscale: stereotyped thinking; and items 1, 9, and 12 in general psychopathology subscale: somatic concern, unusual thought content, lack of judgment, and insight. Higher scores indicate worsening.
Time Frame: Change from baseline to Week 6 or the last post-randomization assessment during double-blind treatment
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Paliperidone Extended-Release (ER)
Number analyzed (Participants) | 93 | 211
points on a scale | -3.3 (5.8) | -6.0 (6.9)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended-Release (ER); Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Means Difference = -2.7, 95% CI [-4.2 to -1.1], Standard Error of Mean 0.8 — Paliperidone Extended Release (ER) - Placebo on the Change Scores

7. Secondary Outcome: Positive and Negative Symptoms of Schizophrenia (PANSS) Negative Factor Score - Change From Baseline to Week 6 Last Observation Carried Forward (LOCF) End Point.
Description: Negative PANSS Factor Score (range 7-49): Sum of scores for items 1, 2, 3, 4, and 6 in negative subscale: blunted affect, emotional withdrawal, poor rapport, passive social withdrawal, lack of spontaneity; and items 7 and 16 in general psychopathology subscale: motor retardation, and active social avoidance. Higher scores indicate worsening.
Time Frame: Change from baseline to Week 6 or the last post-randomization assessment during double-blind treatment
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Paliperidone Extended-Release (ER)
Number analyzed (Participants) | 93 | 211
points on a scale | -1.1 (5.7) | -3.1 (5.2)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended-Release (ER); Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Means Difference = -2.1, 95% CI [-3.3 to -0.9], Standard Error of Mean 0.6 — Paliperidone Extended Release (ER) - Placebo on the Change Scores

8. Secondary Outcome: Positive and Negative Symptoms of Schizophrenia (PANSS) Disorganized Thought Factor Score - Change From Baseline to Week 6 Last Observation Carried Forward (LOCF) End Point.
Description: Disorganized Thoughts PANSS Factor Score (range 7-49): Sum of scores for item 2 in positive subscale:Conceptual disorganization; item 5 in negative subscale:difficulty in abstract thinking; and items 5, 10, 11, 13, and 15 in general psychopathology subscale: mannerisms/posturing, disorientation, poor attention, disturbance of volition, and preoccupation. Higher scores indicate worsening.
Time Frame: Change from baseline to Week 6 or the last post-randomization assessment during double-blind treatment
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Paliperidone Extended-Release (ER)
Number analyzed (Participants) | 93 | 211
points on a scale | -1.4 (4.3) | -3.3 (4.5)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended-Release (ER); Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Means Difference = -1.9, 95% CI [-2.9 to -0.9], Standard Error of Mean 0.5 — Paliperidone Extended Release (ER) - Placebo on the Change Scores

9. Secondary Outcome: Positive and Negative Symptoms of Schizophrenia (PANSS) Uncontrolled Hostility/Excitement Factor Score - Change From Baseline to Week 6 Last Observation Carried Forward (LOCF) End Point.
Description: Uncontrolled Hostility/Excitement PANSS Factor Score (range 4-28): Sum of scores for items 4 and 7 in positive subscale: excitement, hostility; and items 8 and 14 in general psychopathology subscale: uncooperativeness, and poor impulse control. Higher scores indicate worsening.
Time Frame: Change from baseline to Week 6 or the last post-randomization assessment during double-blind treatment
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Paliperidone Extended-Release (ER)
Number analyzed (Participants) | 93 | 211
points on a scale | -2.7 (4.2) | -4.3 (4.4)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended-Release (ER); Test type: Superiority or Other; p = 0.001, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Means Difference = -1.6, 95% CI [-2.6 to -0.6], Standard Error of Mean 0.5 — Paliperidone Extended Release (ER) - Placebo on the Change Scores

10. Secondary Outcome: Positive and Negative Symptoms of Schizophrenia (PANSS) Anxiety/Depression Factor Score - Change From Baseline to Week 6 Last Observation Carried Forward (LOCF) End Point.
Description: Anxiety/Depression PANSS Factor Score (range 4-28): Sum of scores for items 2, 3, 4, and 6 in general psychopathology subscale: Anxiety, Guilt feelings, Tension, Depression. Higher scores indicate worsening.
Time Frame: Change from baseline to Week 6 or the last post-randomization assessment during double-blind treatment
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Paliperidone Extended-Release (ER)
Number analyzed (Participants) | 93 | 211
points on a scale | -2.3 (3.6) | -3.3 (3.7)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended-Release (ER); Test type: Superiority or Other; p = 0.016, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Means Difference = -1.0, 95% CI [-1.8 to -0.2], Standard Error of Mean 0.4 — Paliperidone Extended Release (ER) - Placebo on the Change Scores

11. Secondary Outcome: Clinical Global Impression (CGI-S) - Severity for Schizoaffective Disorder Score at Baseline
Description: The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a subject. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill subjects". Higher scores indicate worsening.
Time Frame: Baseline
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Paliperidone Extended-Release (ER)
Number analyzed (Participants) | 93 | 211
points on a scale | 4.6 (0.6) | 4.6 (0.7)

12. Secondary Outcome: Clinical Global Impression (CGI-S) - Severity for Schizoaffective Disorder - Change From Baseline to Week 6 Last Observation Carried Forward (LOCF) End Point.
Description: as for outcome 11
Time Frame: Change from baseline to Week 6 or the last post-randomization assessment during double-blind treatment
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Paliperidone Extended-Release (ER)
Number analyzed (Participants) | 93 | 211
points on a scale | -0.7 (1.2) | -1.2 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended-Release (ER); Test type: Superiority or Other; p = 0.002, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Means Difference = -0.5, 95% CI [-0.7 to -0.2], Standard Error of Mean 0.1 — Paliperidone Extended Release (ER) - Placebo on the Change Scores

13. Secondary Outcome: Clinical Global Impression (CGI-C) - Change for Schizoaffective Disorder
Description: The CGI-C rating scale is a 7 point global assessment that measures the clinician's impression of the change occurring in the illness over a course of treatment, relative to baseline. A rating of 4 is equivalent to "No change". Ratings of <4 are equivalent to "improvement" and ratings of > 4 are equivalent to "worsening". Higher scores indicate worsening.
Time Frame: Week 6 or the last post-randomization assessment during double-blind treatment
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Paliperidone Extended-Release (ER)
Number analyzed (Participants) | 93 | 211
points on a scale | 3.4 (1.5) | 2.8 (1.3)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended-Release (ER); Test type: Superiority or Other; p < 0.001, ANOVA; P-value is from an ANOVA model with fixed effects for treatment, concomitant medication stratum, and country; LS Means Difference = -0.6, 95% CI [-0.9 to -0.3], Standard Error of Mean 0.2

14. Secondary Outcome: Participants With Response
Description: Response is defined as a 30% or more reduction from baseline PANSS total score and CGI-C score of <= 2 (CGI-C-SCA: Clinical Global Impression of Change for Schizoaffective Disorder).
Time Frame: Week 6 LOCF End Point
Population: Intent-to-Treat
Measure: Number; unit: participants
Arm/Group | Placebo | Paliperidone Extended-Release (ER)
Number analyzed (Participants) | 93 | 211
participants | 26 | 85
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended-Release (ER); Test type: Superiority or Other; p = 0.046, Cochran-Mantel-Haenszel; P-value based on Cochran-Mantel-Haenszel (CMH) chi-square test with modified ridit scores, stratified by concomitant medication stratum, and country

15. Other Pre Specified Outcome: Baseline Hamilton Rating Scale for Depression (HAM-D-21) With Baseline HAM-D-21 Total Score >= 16
Description: Clinician-rated scale that evaluates depressed mood as well as the vegetative and cognitive symptoms of depression. The items are rated on either a 5-point (0 to 4) or a 3-point (0 to 2) scale. The 5-point scale uses a rating of 0 (absent), 1 (doubtful to mild), 2 (mild to moderate), 3 (moderate to severe), and 4 (very severe). Higher scores indicate worsening. The responses are summed to yield the HAM-D-21 score that ranges from 0-63.
Time Frame: Baseline
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Paliperidone Extended-Release (ER)
Number analyzed (Participants) | 65 | 145
points on a scale | 24.6 (5.3) | 24.6 (6.0)

16. Other Pre Specified Outcome: Hamilton Rating Scale for Depression (HAM-D-21) With Baseline HAM-D-21 Total Score >= 16 - Change From Baseline to Week 6 Last Observation Carried Forward (LOCF) End Point.
Description: as for outcome 15
Time Frame: Change from baseline to Week 6 or the last post-randomization assessment during double-blind treatment
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Paliperidone Extended-Release (ER)
Number analyzed (Participants) | 65 | 145
points on a scale | -6.2 (8.6) | -10.2 (8.7)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended-Release (ER); Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Means Difference = -4.1, 95% CI [-6.4 to -1.7], Standard Error of Mean 1.2 — Paliperidone Extended Release (ER) - Placebo on the Change Scores

17. Other Pre Specified Outcome: Baseline Young Mania Rating Scale (YMRS) With Baseline YMRS Total Score >= 16
Description: 11-item scale (elevated mood, increased motor activity, sexual interest, sleep, irritability, speech [rate/amount], language-thought disorder, content, disruptive-aggressive behaviors, appearance, and insight) based on subject's report of his or her condition and clinician's behavioral observations during the interview, with emphasis on the latter. Higher scores indicate worsening. The responses are summed to yield the YMRS total score, which ranges from 0 to 60.
Time Frame: Baseline
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Paliperidone Extended-Release (ER)
Number analyzed (Participants) | 70 | 161
points on a scale | 26.9 (8.1) | 27.5 (7.0)

18. Other Pre Specified Outcome: Young Mania Rating Scale (YMRS) With Baseline YMRS Total Score >= 16 - Change From Baseline to Week 6 Last Observation Carried Forward (LOCF) End Point.
Description: as for outcome 17
Time Frame: Change from baseline to Week 6 or the last post-randomization assessment during double-blind treatment
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Paliperidone Extended-Release (ER)
Number analyzed (Participants) | 70 | 161
points on a scale | -5.7 (10.0) | -10.6 (10.8)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended-Release (ER); Test type: Superiority or Other; p = 0.001, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Means Difference = -4.8, 95% CI [-7.7 to -2.0], Standard Error of Mean 1.5 — Paliperidone Extended Release (ER) - Placebo on the Change Scores

ADVERSE EVENTS:
Description: Safety Population. Safety population for Placebo is 95 subjects and for PALI ER is 214 subjects.
Arm/Group | Placebo | Paliperidone Extended-Release (ER)
Serious Adverse Events (participants affected / at risk) | 8/95 | 11/214
Other Adverse Events (participants affected / at risk) | 22/95 | 66/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=95) | Paliperidone Extended-Release (ER) (N=214)
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Mania (Psychiatric disorders) | 2 | 3
Persecutory delusion (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 2 | 0
Schizoaffective disorder (Psychiatric disorders) | 3 | 5
Suicidal ideation (Psychiatric disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=95) | Paliperidone Extended-Release (ER) (N=214)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 12 (13)
Akathisia (Nervous system disorders) | 1 (1) | 13 (14)
Dizziness (Nervous system disorders) | 5 (5) | 18 (19)
Headache (Nervous system disorders) | 12 (15) | 32 (38)
Insomnia (Psychiatric disorders) | 5 (7) | 14 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days